CLINICAL TRIAL: NCT01684696
Title: Virtual Intervention for Lung Cancer
Acronym: VILC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to secure funding
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 12-09184; (pC ID): 237290 (Other Grant/Funding Number: TRDRP 21XT-0063)
Record Dates: First submitted 2012-09-05; First posted 2012-09-13 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Lung Neoplasms
Keywords: Lung cancer; stigma; virtual intervention; mHealth
MeSH Terms: conditions — Lung Neoplasms; Social Stigma | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mHealth TLC (Experimental): The mhealth TLC group will meet with a nurse before each of 4 clinician visits and use the mHealth TLC on an iPad with an interactive 3-dimensional intervention that allows individuals to experience virtual visits with their clinicians. Key aspects of mHealthTLC include informational videos about lung cancer and LCS. Blame and self-blame will be addressed, information about the role of addiction, social/cultural factors, and tobacco industry influence on smoking behaviors will be highlighted. Patients will experience practiced interaction in ever increasing complex situations with avatars (i.e., receptionist, medical assistant, and clinician). A "virtual coach" will accompany the patient through the virtual visit and will provide information and coaching (as needed).
  Interventions: Behavioral: Virtual experience
- Attention Control (Active Comparator): Attention control group (ACG) - Patients assigned to the ACG will meet with a nurse and receive only the informational videos on an iPad before 4 clinician visits with assessments after each clinician visit. An effort will be made to match the intervention condition on salience, credibility, and contact time.
  Interventions: Behavioral: Videos

INTERVENTIONS:
Behavioral: Virtual experience
  Arms: mHealth TLC
Behavioral: Videos
  Arms: Attention Control

SUMMARY:
Lung cancer is the leading cause of cancer death in both men and women. Lung cancer is unique because of racial disparity, persistent mortality rate, and social stigma. Lung cancer stigma (LCS) and difficult patient-clinician communication may be an underlying factor in health disparities in lung cancer. The purpose of this study is to PILOT test, in a diverse sample of lung cancer patients the effectiveness of the mHealth Tool for Lung Cancer patients (mHealthTLC), an interactive, immersive 3-dimensional iPad application that allows individuals to experience first person virtual visits with their clinicians, to improve patient-clinician communication, decrease LCS, and promote optimal self-management. The study hypotheses are that patients who receive the mHealth TLC will improve their ability to communicate effectively with their clinicians and will report decreased stigma related to their lung cancer diagnosis compared to the attention control group.

DETAILED DESCRIPTION:
This is a two arm experimental design PILOT test of the mHealth Tool for Lung Cancer patients (mHealthTLC) an intervention to improve patient-clinician communication, decrease lung cancer stigma, and decrease lung cancer symptom scores. Patients will be assigned to either the mHealth TLC group or the Attention Control Group (ACG). Interventions in both groups will be delivered online or by iPad in a research office in the clinician's building prior to each visit. Assessments will be done immediately after each visit in the same research room. Intervention and assessment pre-visit is expected to take less than one hour, the intervention is expected to take 30mins, and post assessment is expected to take 30 minutes. A follow-up assessment will be done at 3 months from enrollment.

mhealth TLC group will meet with a nurse just before each of 4 clinician visits and use the mHealth TLC on an iPad with an interactive, immersive 3-dimensional (3-D) intervention that allows individuals to experience virtual visits with their clinicians. The mHealth TLC provides engagement and experiential learning by delivering important information about symptom management and provides the opportunity to practice a new communication strategy in ever increasing complex situations with a virtual coach, receptionist, assistant, and clinician.During the mHealthTLC the patient will enter a virtual clinic office, travel through the different aspects of a typical clinic visit, and interact with office staff and clinicians that are represented by avatars. The avatars will be designed to reflect ethnic and cultural diversity. First person is the preferred format for health teaching because the patient is active as self and not represented as an avatar. The first person vantage point facilitates the immersion and immediacy of the experience. Key aspects of mHealthTLC include informational videos about lung cancer (i.e. etiology, diagnosis, treatment, symptoms) and LCS. Blame and self-blame will be addressed, information about the role of addiction, social/cultural factors, and tobacco industry influence on smoking behaviors will be highlighted. Information and training will be provided and patients will be able to experience practiced interaction in ever increasing complex situations with avatars (i.e., receptionist, medical assistant, and clinician). A "virtual coach" will accompany the patient through the virtual visit and will provide information and coaching (as needed). The advantages to adding a virtual coach or avatar include the availability of an always-live agent and the capability of customizing the coach to represent an ideal social model for a particular user or group of users.Flexibility exists in how to design not only how the coach will appear but also how the coach will sound - with an appropriate voice and engaging non-verbal communication). This approach contributes to cultural and ethnic sensitivity. As the patient attempts to communicate and receive information appropriate for a self-management plan, they will receive "points" for successful communication. A cumulative score and explanation will be given at the end of the virtual visit. During the visit the participant will identify specific topics and questions that they want to address during their visit with their real clinician; they will receive a printout of their priority questions that they can take into the visit with their real clinician. The research nurse will review the score, the priority questions, and the overall virtual experience. Virtual environments for learning are sufficiently promising that further investment and development of this type of research is warranted.

Attention control group (ACG)- Patients assigned to the ACG will meet with a nurse and receive the informational videos from the mHealth TLC on an iPad before 4 clinician visits with assessments after each clinician visit. An effort will be made to match the intervention condition on salience, credibility, and contact time.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are >21 years old with a diagnosis of lung cancer (any type or stage), able to read and write English at 5th grade level, able to sign an IRB approved consent form, and expects to have 4 visits with the same clinician in the next 2 months.

Exclusion Criteria:

* Unable to understand or tolerate the battery of questionnaires due to physical or mental health issues (i.e., dementia, active psychosis).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Patient-clinician communication scores | 3 months
  The Medical Communication Competence Scale (MCCS) measures patients' perceptions of their competence to effectively communicate. The Patients' Self-Competence Subscale of the MCCS has 16-items with a 5 point Likert-type scaling of 5 (important) to 1 (unimportant). Higher scores indicate greater perceived self-competence. The Quality of Physician-Patient Interaction (QQPPI) measures distinct domains that establish a high quality clinician-provider interaction (i.e.,information exchange, patient involvement, and sharing in the decision making process). Fourteen items are summed to yield a total score; higher scores indicate increased quality of communication as perceived by the patient.
Perceived lung cancer stigma | 3 months
  The Cataldo Lung Cancer Stigma Scale (CLCSS) will be used to assess stigma. The CLCSS is a 31 item measure with each item rated on a 4-point Likert-type scale (strongly disagree to strongly agree). Higher values indicate higher levels of LCS.The CLCSS was found to be a reliable and valid measure with a diverse sample of people with lung cancer. Construct validity was supported by expected relationships with related constructs: self-esteem, depression, social support, and social conflict. The total scale Cronbach alpha coefficient was 0.96, the Cronbach alphas for the four subscales were: stigma/shame, 0.96; social isolation, 0.95; discrimination, 0.92; and smoking 0.76.

SECONDARY OUTCOMES:
Lung Cancer symptoms | 3 months
  Lung Cancer Symptoms - Lung Cancer Symptom Scale (LCSS) measures the physical and functional dimensions of persons with lung cancer. The scale has 9 items: six measuring major symptoms for lung cancer (appetite loss, fatigue, cough, dyspnea, hemoptysis, pain) and three summary items related to total symptoms. The item scale is 0 (best) and 100 (worst). An average of all 9 items is the total score.
Depression | 3 months
  Depression - Center for Epidemiologic Studies-Depression (CES-D) is a 20-item scale that is widely used for self-ratings of depression in clinical populations, including people with cancer.
Quality of Life (QOL) | 3 months
  QOL - The QOL Inventory is a 33-item instrument that measures four dimensions of QOL in cancer patients (i.e., symptoms, social concerns, psychological well-being, and physical well being).

CONTACTS AND LOCATIONS:
Overall Officials: Janine Cataldo, PhD, Principal Investigator — UCSF Department of Physiological Nursing
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States